CLINICAL TRIAL: NCT02607774
Title: An Open-label, Single Sequence Crossover, Study Investigating the Influence of Secukinumab Treatment on the Pharmacokinetics of Midazolam as a CYP3A4 Substrate in Patients With Moderate to Severe Plaque Psoriasis
Brief Title: Investigate Effect of Secukinumab on the PK of Midazolam in Patients With Mod to Sev Plaque Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CAIN457A2110
Record Dates: First submitted 2015-11-03; First posted 2015-11-18 (Estimated); Last update posted 2020-12-11 (Actual); Status verified 2019-03

CONDITIONS: Moderate to Severe Plaque Psoriasis
Keywords: Plaque psoriasis; disease-drug-drug-interaction; midazolam; secukinumab
MeSH Terms: interventions — Midazolam; secukinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Secukinumab (Experimental): Secukinumab over 24 weeks
  Interventions: Drug: Midazolam; Drug: AIN457

INTERVENTIONS:
Drug: Midazolam — midazolam administered to all patients Days -7, 1 and 35.
Drug: AIN457 — secukinumab administered at Weeks 0, 1, 2, 3, 4, 8, 12, 16, 20 and 24
  Other Names: Secukinumab

SUMMARY:
To determine whether secukinumab can alter the activity of cytochrome P450 (CYP) 3A4 using midazolam as probe substrate in patients with moderate-to-severe plaque psoriasis.

DETAILED DESCRIPTION:
This will be an open-label, confirmatory study investigating potential disease-drug-drug interaction of secukinumab and midazolam in male and female patients with moderate-to-severe plaque psoriasis. A total of approximately 25 patients are required to obtain at least 20 completers in the study Patients who meet the eligibility criteria at screening, will have a baseline assessment day (within 1 week prior to the start of secukinumab) during which a full midazolam PK profile after a single oral dose of 5 mg will be assessed by collecting blood over the 12 hour postdose period.

On Day 1 (Week 0), Day 8 (Week 1), Day 15 (Week 2), Day 22 (Week 3) and Day 29 (Week 4) patients will receive 300 mg s.c. secukinumab (2 injections of 150 mg s.c.). On Day 8 and on Day 36 (Week 5), patients will receive additional single doses of 5 mg oral midazolam (total of 3 single doses). The midazolam PK profile will be assessed over the 12 hour postdose period.

On those days when midazolam PK profiles are assessed, samples will be collected and analyzed for circulating IL-6, inflammatory panel (collected at screening, baseline and pre-dose Day 1 only), total IL-17A (after following initiation of secukinumab treatment), hsCRP and for 4-beta-hydroxycholesterol (exploratory endogenous phenotyping marker of CYP3A activity).

There will be an extended treatment period during which patients will receive secukinumab 300 mg s.c. at Weeks 8, 12, 16, 20 and 24.

Then there will be a follow-up period of 12 weeks following the last dose administered at Week 24. Visits will be at Weeks 28, 32 and 36.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe plaque psoriasis as defined at baseline by: PASI score of 12 or greater and IGA mod 2011 score of 3 or greater (based on a scale of 0 - 4) and Body Surface Area (BSA) affected by plaque-type psoriasis of 10% or greater.
* Chronic plaque-type psoriasis considered inadequately controlled by: topical treatment and/or; phototherapy and/or previous systemic therapy
* Men or women at least 18 years of age or older at time of screening.

Exclusion Criteria:

* Forms of psoriasis other than chronic plaque-type
* Pregnant or nursing (lactating) women,
* History of an ongoing, chronic or recurrent infectious disease, or evidence of tuberculosis infection.
* Subjects with known history of hypersensitivity to midazolam

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-12-17 (Actual); Primary Completion 2016-12-20 (Actual); Study Completion 2016-12-20 (Actual)

PRIMARY OUTCOMES:
Cmax (maximum plasma) concentration | Days -7, 8 and 36
AUC0-12 (area under the plasma concentration-time curve from time zero to time 12 hours ) | Days -7, 8 and 36
AUClast (area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration) | Days -7, 8 and 36
AUCinf (area under the plasma concentration-time curve from time zero to infinity) | Days -7, 8 and 36

SECONDARY OUTCOMES:
safety and tolerability (including; Blood pressure,Pulse Rate,AEs/SAEs, Blood chemistry, Hematology, ECGs and physical exam | Throughout the entire trial; beginning at screening through Day 253 (end of trial)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Hot Springs, Arkansas
  - Novartis Investigative Site, Fair Lawn, New Jersey
  - Novartis Investigative Site, Verona, New Jersey
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Webster, Texas
  - Novartis Investigative Site, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=203
- See also: Results for CAIN457A2110 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=16935